CLINICAL TRIAL: NCT02862483
Title: The Efficacy and Safety of the Combination of Tamsulosin and Tadalafil in Men With Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia and Erectile Dysfunction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-TATA-301
Record Dates: First submitted 2016-07-22; First posted 2016-08-11 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Benign Prostatic Hyperplasia; Erectile Dysfunction
MeSH Terms: conditions — Prostatic Hyperplasia; Erectile Dysfunction | interventions — Tamsulosin; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Tamsulosin 0.2mg and Tadalafil 5mg
  Interventions: Drug: Tamsulosin 0.2mg; Drug: Tadalafil 5mg
- Comparator (Active Comparator): placebo for Tamsulosin 0.2mg and Tadalafil 5mg
  Interventions: Drug: Tadalafil 5mg; Drug: Placebo for Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin 0.2mg
  Arms: Experimental
Drug: Tadalafil 5mg
Drug: Placebo for Tamsulosin
  Arms: Comparator

SUMMARY:
The efficacy and safety of the combination of tamsulosin and tadalafil in men with lower urinary tract symptoms due to benign prostatic hyperplasia and Erectile Dysfunction: a randomized, double blinded, parallel design, active controlled, multi-center, phase 3 clinical trial

ELIGIBILITY:
Inclusion Criteria:

Visit1

* Male aged 45 years old or older
* Subjects who have PSA ≤ 4.0 ng/mL Visit2
* Subjects who have Total IPSS score ≥ 13
* Subjects who have IIEF-EF domain ≤ 24 and each point below 3 in question 3 and 4

Exclusion Criteria:

* Subjects who have hypersensitivity to investigational product or sulfa medications

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The change of total IPSS(International prostate symptom score) | From baseline at week 12
The change of IIEF-EF(International Index of Erectile Function sum of questions-Erectile function) domain | From baseline at week 12

SECONDARY OUTCOMES:
The change of total IPSS(International prostate symptom score) | From baseline at week 4,8
The change of total IPSS(International prostate symptom score) sub score (storage, voiding) | From baseline at week 4,8 and 12
The change of IPSS(International prostate symptom score) QoL(Quality of Life) | From baseline at week 4,8 and 12
The change of Qmax(maximum urinary flow rate) | From baseline at week 4,8 and 12
The change of PVR(Post Void Residual Volume) | From baseline at week 4,8 and 12
PGIC(Patient Global Impression of change) score | At week 12
CGIC(Clinician Global Impression of change) score | At week 12
The change of IIEF (International Index of Erectile Function sum of questions) total score | From baseline at week 4,8 and 12
The change of IIEF-IS(International Index of Erectile Function sum of questions-Intercourse satisfaction) domain score measured by IIEF question number 6~8 | From baseline at week 4,8 and 12
The change of OS(Overall satisfaction) domain score measured by IIEF question number13 and 14 | From baseline at week 4,8 and 12
The change of OF(Orgasmic function) domain score measured by IIEF question number 9 and 10) | From baseline at week 4,8 and 12
The change of IIEF-EF domain(International Index of Erectile Function sum of questions-Erectile function) score measured by IIEF question number 1~5 and 15 | From baseline at week 4,8
The change of IIEF(International Index of Erectile Function) score about questions number 3 and 4 | From baseline at week 12
The percentage of patients who have more than 4 point about IIEF questions number 3 and 4 | From baseline at week 12
The percentage of patients who have increased score about IIEF questions number 3 and 4(at least 1 point) compared to the baseline | From baseline at week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic university of korea, Seoul ST. Mary's Hospital., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No